CLINICAL TRIAL: NCT01933204
Title: Acupuncture for Relieving Perimenopausal Symptoms: a Randomised Controlled Trial
Brief Title: Acupuncture for Relieving Perimenopausal Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Chengdu First People's Hospital (Other); Chengdu PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012BAI24B01
Record Dates: First submitted 2013-08-09; First posted 2013-09-02 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Perimenopause
Keywords: perimenopause; hot flash; palpitation
MeSH Terms: conditions — Hot Flashes | interventions — Acupuncture Therapy; estradiol valerate, cyproterone acetate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Using basic points combined with additional points. Basic points are fixed, while additional points will be selected from a list of points categorized by syndrome differentiation.
  Interventions: Other: Acupuncture
- Climen 21 Tablets (Active Comparator): COMPOSITION 11 white tablets each containing estradiol-17-valerate 2 mg, plus 10 pink tablets each containing estradiol-17-valerate 2 mg and cyproterone acetate 1 mg.
  Interventions: Drug: Climen 21 Tablets

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a collection of procedures involving penetration of the skin with needles to stimulate certain points on the body. In its classical form it is a characteristic component of traditional Chinese medicine (TCM), a form of alternative medicine, and one of the oldest healing practices in the world.
  Arms: Acupuncture
Drug: Climen 21 Tablets — Climen Tablets are commonly used for menopausal symptoms
  Other Names: Climen Tablets
  Arms: Climen 21 Tablets

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective for relieving perimenopausal symptoms.

DETAILED DESCRIPTION:
* A randomised controlled trial with superiority design
* A total of 220 participants will be included in 3 centers
* 2 arms: acupuncture group and Climen® group

ELIGIBILITY:
Inclusion Criteria:

* Participants who complained of irregular menstrual cycle in the past 12 months, with a forward or postpone of a cycle more 7 days. At least 2 cycles were missing during the past 12 months, or reported menopause for at least 60 days.
* Reported relative perimenopausal symptoms, e.g., hot flash, insomnia, migraine, easy irritation, etc.
* Age 40-50 years.
* Not accompanied with conditions that are needed for hormone therapy, e.g., menopause after surgery, active osteoporosis.
* Willing to participate and signing the inform consent.

Exclusion Criteria:

* Had a regular menopausal cycle 3 months before this trial.
* Taking estrogen, selective serotonin reuptake inhibitor(SSRI), soy isoflavone, progesterone, Vitamin E or black cohosh in the 4 weeks before inclusion.
* receiving chemoradiotherapy.
* Agnogenic vaginal bleeding.
* Coagulation defeats, or taking anticoagulant drugs, such as warfarin, heparin, etc.
* Dermal diseases, e.g., eczema, psoriasis.
* Liver or kidney failure.
* Uncontrollable hypertension, diabetes, or thyroid diseases.
* With diabetic neuropathy, malignant cancer and mental diseases (including depression).
* Intend to gestation, in gestation period or lactation period.
* Using sedative or antianxiety drugs.
* With smoking or intemperance problems.
* Using cardiac pacemaker, or joint prosthesis.
* Low compliance.
* Benign tumor in breast.
* Family history of breast cancer.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale | 12 weeks after randomization
  The scale was developed and validated over the years from a research network of many institutions such as Organon Germany, Infratest Munich, Universities of Muenster and Berlin,the Berlin Center for Epidemiology and Health Research, etc. It is a scale consisted of 11 items, ranging from no symptoms to very severe symptoms.

SECONDARY OUTCOMES:
Menopausal Specific Quality of Life Questionnaire | asessed 0, 6, 12, 24, 36 weeks after randomization
  The Menopausal Specific Quality of Life Questionnaire (MENQOL) is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29).
Average hot flash score during 24 hours | 0, 12, 24, 36 weeks after randomization
Level of Estradiol in serum | 0, 12, 24 weeks after randomization
Level of follicle stimulating hormone in serum | 0, 12, 24 weeks after randomization
Level of luteinizing hormone in serum | 0, 12, 24 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ying Li, MD, PhD, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - First affiliated hospital of Chengdu University of TCM, Chengdu, Sichuan

REFERENCES:
- [Derived] Li Y, Zheng H, Zheng Q, Zhao L, Qin E, Wang Y, Zeng Q, Zheng H, Zhao Y, Sun W, Zhang X, Liu Z, Liu B. Use acupuncture to relieve perimenopausal syndrome: study protocol of a randomized controlled trial. Trials. 2014 May 30;15:198. doi: 10.1186/1745-6215-15-198. PMID 24886348